CLINICAL TRIAL: NCT01581294
Title: Long-term Safety and Effectiveness of Disease Modifying Therapies in Inflammatory Arthropathies: a Multicentre, Phase IV, Longitudinal Observational Study
Brief Title: The Norwegian Antirheumatic Drug Register
Acronym: NOR-DMARD
Status: Recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University Hospital of North Norway (Other); St. Olavs Hospital (Other); Lillehammer Hospital for Rheumatic Diseases (Other); Vestre Viken Hospital Trust (Other); Helse Forde (Other)
Responsible Party: Principal Investigator, Tore K Kvien, Principal Investigator, Diakonhjemmet Hospital
Other Study IDs: DIA 2011-1
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Inflammatory Joint Diseases
Keywords: Rheumatoid arthritis; Psoriatic arthritis; Ankylosing spondylitis; Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples (including serum, plasma and full blood) for biomarker or DNA/RNA discovery and validation will be collected and stored in a freezer at -70 C at visits at baseline and at the 3-month assessment.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
NOR-DMARD is a register-based longitudinal observational study of which the main objectives are to study the effectiveness of treatment of inflammatory joint diseases with biological disease modifying anti-rheumatic drugs (DMARDs) in clinical practice, by measuring disease activity, health related quality of life, function and joint damage, and to study the long-term safety of such treatment. Other objectives include the assessment of cost-effectiveness of treatment, to identify and and validate clinical, genetic and immunological predictors of efficacy and adverse events, to assess the impact of treatment with biological DMARDs on work participation and work productivity, to investigate different strategies for use of biological DMARDs, to assess the performance of different outcome measures, and to ensure a systematic and timely follow-up of patients treated with biological DMARDs.

DETAILED DESCRIPTION:
This study is a modification, and an extension, of the NOR-DMARD study that was conducted in 5 Norwegian rheumatology departments in the period 2000-2012. The study includes a structured follow-up with study visits at baseline (start of biological drug) and after 3, 6, 12 months and every 12 months thereafter. Each study visit includes clinical assessment, patient-reported outcomes and measurement of acute-phase reactants. The data collection also includes blood samples for biobank at baseline and 3 months. Serious adverse events data will be systematically recorded, but other adverse events can also be retrieved by linkage to other registers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, spondyloarthritis, adult juvenile idiopathic arthritis, undifferentiated arthritis, or any other inflammatory arthritis
* Clinical indication to start a new treatment with a biological disease modifying anti-rheumatic drug or a kinase inhibitor

Exclusion Criteria:

* Unwillingness or unability to give written informed consent
* Psychiatric or mental disorders, alcohol abuse or other abuse of substances, language barriers or other factors which makes adherence to the study protocol impossible
* Participation in blinded RCTs or other studies incompatible with the NOR-DMARD study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with inflammatory arthropathies starting a new treatment with a biological disease modifying anti-rheumatic drug
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2012-04; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

SECONDARY OUTCOMES:
Disease Activity Score-28 (DAS28) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
American College of Rheumatology (ACR) responses (ACR20, ACR50, ACR70) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Simplified Disease Activity Index (SDAI) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) remission | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Assessments of Spondyloarthritis International Society (ASAS) responses (ASAS20, ASAS40) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Modified Health Assessment Questionnaire (MHAQ) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Rheumatoid Arthritis Impact of Disease (RAID) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Work Productivity and Activity Impairment (WPAI) Questionnaire | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
EuroQol 5-dimensions (EQ-5D) questionnaire | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
  Utility instrument
28-Swollen joint count | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
28-Tender joint count | All follow-up visits
Erythrocyte Sedimentation Rate (ESR) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
C-Reactive Protein (CRP) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months
Sharp/van der Heijde score | 12, 24, 36, 48, 60 months
  Radiographic progression
Number of participants with adverse events | 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120 months
Clinical Disease Activity Index (CDAI) | 3, 6, 9, 12, 18, 24, 36, 48, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Tore K Kvien, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (6):
- Norway (6):
  - Vestre Viken HF Drammen Hospital, Drammen, Buskerud
  - Lillehammer Hospital for Rheumatic Diseases, Lillehammer, Oppland
  - Førde Hospital, Førde, Sogn Og Fjordane
  - St. Olavs Hospital, Trondheim, Sør-Trøndelag
  - University Hospital of Northern Norway, Tromsø, Troms
  - Diakonhjemmet Hospital, Oslo

REFERENCES:
- [Derived] Mielnik P, Sexton J, Lie E, Bakland G, Loli LP, Kristianslund EK, Rodevand E, Lexberg AS, Kvien TK. Does Older Age have an Impact on Rituximab Efficacy and Safety? Results from the NOR-DMARD Register. Drugs Aging. 2020 Aug;37(8):617-626. doi: 10.1007/s40266-020-00782-x. PMID 32648248
- [Derived] Gehin JE, Goll GL, Warren DJ, Syversen SW, Sexton J, Strand EK, Kvien TK, Bolstad N, Lie E. Associations between certolizumab pegol serum levels, anti-drug antibodies and treatment response in patients with inflammatory joint diseases: data from the NOR-DMARD study. Arthritis Res Ther. 2019 Nov 29;21(1):256. doi: 10.1186/s13075-019-2009-5. PMID 31783773
- [Derived] Olsen IC, Lie E, Vasilescu R, Wallenstein G, Strengholt S, Kvien TK. Assessments of the unmet need in the management of patients with rheumatoid arthritis: analyses from the NOR-DMARD registry. Rheumatology (Oxford). 2019 Mar 1;58(3):481-491. doi: 10.1093/rheumatology/key338. PMID 30508189